CLINICAL TRIAL: NCT05360628
Title: A Phase I, Randomized, Open-label Study to Evaluate the Potential Pharmacokinetic Interactions Between D-0120 and Allopurinol in Healthy Adult Subjects
Brief Title: Evaluation of PK and Safety of D-0120 and Allopurinol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D0120-104
Record Dates: First submitted 2021-11-01; First posted 2022-05-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Allopurinol

STUDY DESIGN:
Intervention Model Description: D0120 Allopurinol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D-0120 plus Allopurinol (Experimental): D-0120 dosing followed by Allopurinol and combination treatment
  Interventions: Drug: D-0120 in combination with Allopurinol
- Allopurinol plus D-0120 (Experimental): Allopurinol dosing followed by D-0120 and combination treatment
  Interventions: Drug: D-0120 in combination with Allopurinol

INTERVENTIONS:
Drug: D-0120 in combination with Allopurinol — noted above

SUMMARY:
Evaluation of safety and PK interaction between D-0120 and Alopurinol in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 18-55
* Required evaluation by Investigator for screening and enrollment
* Agreement and compliance with the study and follow-up procedures

Exclusion Criteria:

* Significant medical history or current comorbidly determined by the Investigator.
* Pregnant or nursing women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-07-23 (Actual)

PRIMARY OUTCOMES:
Type, incidence, severity and attribution of AEs. | 14 days
  Evaluation of safety between D-0120 and Allopurinol
Plasma concentration of D-0120 and Allopurinol | 14 days
  Evaluation of exposure between D-0120 and Allopurinol

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No